CLINICAL TRIAL: NCT01250795
Title: A Phase 1a/b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Investigate the Safety, Reactogenicity, and Immunogenicity of FhCMB HAI-05, a Recombinant Hemagglutinin (rHA) Vaccine Derived From Influenza A/Indonesia/05/2005 (H5N1), in Healthy Adults 18 to 49 Years
Brief Title: Safety and Immunogenicity Of A Recombinant H5N1 Vaccine In Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fraunhofer, Center for Molecular Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FhCMB HAI-05-001
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Prevention
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 15 ug HAI-05 plus Alhydrogel (Experimental): vaccine
  Interventions: Biological: HAI-05 Influenza Vaccine
- 45 ug HAI-05 plus Alhydrogel (Experimental): vaccine
  Interventions: Biological: HAI-05 Influenza Vaccine
- 90 ug HAI-05 plus Alhydrogel (Experimental): vaccine
  Interventions: Biological: HAI-05 Influenza Vaccine
- 90 ug HAI-05 in saline (Experimental): vaccine
  Interventions: Biological: HAI-05 Influenza Vaccine
- Saline (Placebo Comparator): placebo
  Interventions: Other: Saline

INTERVENTIONS:
Biological: HAI-05 Influenza Vaccine — injection, vaccine, twice every 3 weeks
  Arms: 15 ug HAI-05 plus Alhydrogel; 45 ug HAI-05 plus Alhydrogel; 90 ug HAI-05 in saline; 90 ug HAI-05 plus Alhydrogel
Other: Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to assess the safety, immunogenicity,and tolerability of a H5N1 Vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Subjects accepted for this study must meet the following inclusion criteria:

* Male or female aged 18 to 49 years inclusive
* Able to give written informed consent to participate
* Healthy as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations at baseline
* Females should fulfill one of the following criteria:

  1. At least 1 year post-menopausal
  2. Surgically sterile
  3. Will use oral, implantable, transdermal, or injectable contraceptives for 30 days prior to first vaccination and until 28 days after each vaccination
  4. Willing to abstain from sexual intercourse or use another reliable form of contraception approved by the investigator (e.g., intrauterine device [IUD], female condom, diaphragm with spermicide, cervical cap, use of condom by the sexual partner, or a sterile sexual partner) for study duration and until 28 days after vaccination
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of each dose
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits and to be contacted by telephone throughout the follow-up period

Exclusion Criteria:

Any of the following are cause for exclusion from the study:

* Prior receipt of any influenza vaccine containing H5
* Presence of significant uncontrolled medical or psychiatric illness (acute or chronic); includes institution of new medical or surgical treatment or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed on Day 1 prior to vaccination
* Positive serology for human immunodeficiency virus (HIV 1 or HIV 2), hepatitis B surface antigen (HBsAg). or hepatitis C (HCV)
* Cancer or treatment for cancer within 3 years excluding basal cell carcinoma or squamous cell carcinoma which are allowed
* Presence of any medical condition that may be associated with impaired immune responsiveness, including diabetes mellitus
* Presently receiving (or has a history of receiving) during the preceding 3 month period any medications or other treatments that may adversely affect the immune system, such as allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs; other drugs known to be frequently associated with significant major organ toxicity; or systemic (oral or injectable) corticosteroids (inhaled and topical corticosteroids allowed)
* Receipt or planned administration of a nonstudy vaccine within 30 days prior to vaccination and during the study (Immunization on an emergency basis with Tetanus Toxoids Adsorbed for adult use vaccine-tetanus and diphtheria [Td] or tetanus, diphtheria, and pertussis [Tdap] up to 8 days before or at least 8 days after a dose of study vaccine will be allowed, and administration of study vaccine injection can be delayed if a nonstudy vaccine has been administered and will be given as soon as acceptable [as described above] provided the vaccine is not administered within 2 weeks prior to study enrollment.)
* History of significant allergic reactions (anaphylactic-type reactions, respiratory difficulties, or angioedema) to injected vaccines or to any of the study vaccine components
* History of drug or chemical abuse in the year before the study; positive urine drug screen at screening.
* Receipt of any investigational product or nonregistered drug within the 30 days prior to vaccination or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing study period
* Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the study period
* Donation of blood or blood products within 8 weeks prior to vaccination or at any time during the study
* Acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical examination) with or without fever, or a fever >38ºC orally (Study vaccine can be administered to persons with a minor illness, such as diarrhea, or mild upper respiratory tract infection with or without low-grade fever, and vaccination can be delayed until the subject has recovered.)
* Any condition that, in the opinion of the investigator, might interfere with the primary study objectives or the subject's safety

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
safety | 200 days

SECONDARY OUTCOMES:
immunogenicity | day 43

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Heartland Research Associates, LLC, Wichita, Kansas
  - The Center for Pharmaceutical Research, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided